CLINICAL TRIAL: NCT00917475
Title: Socio-Emotional Development in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Dr. Suh-Fang Jeng, School and Graduate Institute of Physical Therapy, National Taiwan University
Other Study IDs: 200904054R
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Preterm Infants
Keywords: preterm infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants: birth weight<1500 grams and gestational age<30 weeks

SUMMARY:
With advances in medicine and medical technology, premature infants born as early as 24 weeks of gestation and with birth weight less than 1000 grams are surviving today. Preterms are born with immature biological systems. Given their biological vulnerabilities, preterm infants are at risk for a variety of health and developmental problems.

As a group, preterms show developmental delays in physical growth, motor skills, attention, social communicative skills, intelligence, language, academic performance, and later behavior problems. Furthermore, research indicates that preterms are difficult social partners for their parents.

Despite biological insults and relational difficulties, research also shows that the development of premature infants appears to be facilitated by sensitive and responsive parenting. Little attention, however, has been paid to understand the social risks faced by preterm infants.

The proposed research, therefore, is designed to:

1. understand the extent to which neurophysiological risk may affect preterm infants' socioemotional development,
2. explore the role of maternal social support, sociopsychological stress, and perception of infant vulnerability in the socioemotional development of preterm infants varying in biological risk,
3. examine the role of social support in buffering stress in mothers of preterm infants, and
4. evaluate the role of maternal stress, coping, and support in preterm infants' socioemotional development.

This study will include preterm infants recruited from the National Taiwan University Hospital at term and 12 months of corrected age. Infants will be examined for physical growth, neurobehavioral development, and mother and infant interaction at term. The growth measures including weight, height and head circumference will be assessed. Interaction between mother and infant will be investigated by observing the interaction between infants and their mothers in feeding and skin to skin contact conditions. Mothers' psychosocial stress and social support will be obtained via questionnaires.

It is expected that preterm infants' physical growth and neurobehavioral development as well as mothers' psychosocial stress and social support are associated with the quality of mother-infant interaction.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants

Exclusion Criteria:

* significant congenital problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants born prematurely with no significant congenital problems (e.g., cleft palate, cardiac malformations) and their mothers ages 18 to 40.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
quality of mother-infant interaction | term age and 12 months of corrected age

SECONDARY OUTCOMES:
maternal parenting efficacy | term age and 12 months of corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chin Hsu, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan